CLINICAL TRIAL: NCT00341718
Title: The Experiences of Genetics Patients With Visible Differences Who Facilitate Teaching in Genetics Clinics
Brief Title: Experiences of Genetics Patients With Visible Abnormalities Who Facilitate Teaching in Genetics Clinics
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906130; 06-HG-N130
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-03-31

CONDITIONS: Learning
Keywords: Interview; Genetics

SUMMARY:
This study will describe the experience of patients with visible physical abnormalities in the genetics clinic when they are involved in teaching others about their condition. Information from this study may be used to enhance educational experiences in genetics clinics.

Patients 18 years of age and older with a visible physical anomaly who have been seen by a genetics professional in the past 5 years may be eligible for this study.

In a tape-recorded telephone interview, patients are asked about the following:

* Their experiences when visiting the genetics clinic
* The circumstances under which they have been approached to participate in teaching others
* Their perspective on specific teaching behaviors used in genetic consultations, and how this perspective is affected by their perception of their own visible difference
* The benefits and downsides of being involved in teaching others
* The circumstances under which they feel comfortable being approached by genetics providers to help teach others about their condition
* The conditions or circumstances that make some individual teaching experiences better or worse than others

DETAILED DESCRIPTION:
It is common for genetics patients to facilitate teaching of others during the course of their genetics exam. Patient response to serving as a teaching case has been studied only on a limited extent. This study proposes to qualitatively explore the ways in which taking on a teaching role in a genetics clinic is experienced by patients with visible differences.

Qualitative telephone interviews with approximately 30 genetics patients with visible differences will be conducted. The interviews will be semi-structured and an interview guide will be loosely followed. Interviews will be recorded and transcripts of the interviews will be coded for analysis. A typology of common themes will be compiled and reported. Information collected through these interviews will improve understanding of the phenomenon of patients in educator roles, relate experiences to patient expectations and will fill a gap in the published literature. It is additionally hoped that results of this study may inform the development of new recommendations to enhance educational experiences in genetics clinics.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Seen in a genetics clinic or by a genetics professional in the past 5 years.
  2. Self-reported obvious physical difference or deformity.
  3. English speaking.

EXCLUSION CRITERIA:

1. Younger than 18 years.
2. Non-visible or absent physical difference of deformity.
3. Cognitively-impaired or incompetent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-03-29; Study Completion 2007-03-31

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Wright HJ. Patients' attitudes to medical students in general practice. Br Med J. 1974 Mar 2;1(5904):372-6. doi: 10.1136/bmj.1.5904.372. PMID 4819176